CLINICAL TRIAL: NCT06818669
Title: Cardiovascular Risk Reduction for Adults With Food Insecurity Using Structured Incentives (CVD-FIT)
Brief Title: Cardiovascular Risk Reduction for Adults With Food Insecurity Using Structured Incentives
Acronym: CVD-FIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Rebekah Jo Walker, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: R01MD018721 (NIH); 1R01MD018721-01A1 (NIH)
Record Dates: First submitted 2025-02-07; First posted 2025-02-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cardiovascular Diseases
Keywords: Food Insecurity; Financial Incentives
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to CVD-FIT (a multi-component intervention that includes three components: 1) monthly income supplementation; 2) weekly structured incentive for the purchase of healthy food options; and 3) evidence-based telephone delivered CVD risk reduction education and skills training) or enhanced usual care (CVD risk reduction education).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CVD-FIT (Experimental): The structured incentive will include monthly supplemental income plus weekly reimbursement for the purchase of healthy food options. Education for CVD risk reduction will include mailed education and telephone calls with a trained health educator.
  Interventions: Behavioral: CVD-FIT
- Enhanced Usual Care (Active Comparator): Education for CVD risk reduction will include mailed education and telephone calls with a trained health educator.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: CVD-FIT — The structured incentive will include monthly supplemental income plus weekly reimbursement for the purchase of healthy food options. Education for CVD risk reduction will include mailed education and telephone calls with a trained health educator.
  Arms: CVD-FIT
Behavioral: Enhanced Usual Care — Education for CVD risk reduction will include mailed education and telephone calls with a trained health educator.
  Arms: Enhanced Usual Care

SUMMARY:
The overarching aim of this proposal is to test the efficacy and cost-effectiveness of CVD-FIT, a novel, multi-component intervention that includes three components: 1) monthly income supplementation; 2) weekly structured incentive for the purchase of healthy food options; and 3) evidence-based telephone delivered CVD risk reduction education and skills training in African Americans with food insecurity.

DETAILED DESCRIPTION:
Study Overview: 200 African American adults at risk for CVD with food insecurity will be randomized 1:1 to CVD-FIT or enhanced usual care (CVD risk reduction education). Each patient will be followed for 12 months, with study visits at baseline, 3, 6, and 12 months. The primary outcome will be 10-year CVD risk using the Pooled Cohort Equation at 12 months post-randomization while the secondary outcomes will be quality of life at 12 months post-randomization and cost-effectiveness of the CVD-FIT intervention compared to enhanced usual care.

Patient Randomization. A permuted block randomization method will be used to assign subjects to intervention or control. All subjects who are randomized will be entered into the study database and analyzed according to CONSORT guidelines.

Description of the CVD-FIT Intervention: The CVD-FIT intervention will incorporate 1) $100 monthly income supplementation; 2) $50 weekly structured incentive for the purchase of healthy food options; and 3) evidence-based telephone delivered CVD risk reduction education and skills training.

Enhanced Usual Care Control Group: Participants randomized to the enhanced usual care group will receive the same mailed education and health educator delivered education and skills training sessions as the CVD-FIT intervention group.

ELIGIBILITY:
Inclusion Criteria:

* self-report as African American/non-Hispanic Black
* screen positive for food insecurity over the past 12-months using a food insecurity risk tool developed through completion of the research team's current NIH funded R01 (R01MD013826)
* at risk for CVD defined as age ≥40 years and having a clinical diagnosis of diabetes, or hypertension, or hyperlipidemia, or being overweight/obese (defined as a BMI>25), or being a current smoker
* able to communicate in English.

Exclusion Criteria:

* Mental confusion on interview suggesting significant dementia
* Participation in other cardiovascular disease clinical trials
* Alcohol or drug abuse/dependency based on screening using CAGE questionnaire
* Active psychosis or acute mental disorder based on self-report
* Life expectancy <12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
10-Year CVD Risk | baseline, 3-months, 6-months, and 12-months post randomization
  10-year CVD risk will be measured by the Pooled Cohort risk reduction equation recommended for race- and sex- specific risk calculation for African Americans 40 to 79 years of age.
CVD Risk - PREVENT | baseline, 3-months, 6-months, and 12-months post randomization
  CVD Risk will be measured using the PREVENT equation

SECONDARY OUTCOMES:
Physical and Mental Health Related Quality of Life | baseline, 3-months, 6-months, and 12-months post randomization
  Quality of Life will be measured using the SF-12 questionnaire and reported as physical health related and mental health related scores (score ranges from 0 to 100 with higher numbers indicating better quality of life)

CONTACTS AND LOCATIONS:
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared to protect privacy of participants